CLINICAL TRIAL: NCT04698590
Title: Custom Anterior Surfacing of Scleral Lens for Vision Quality Improvement in Patients With Keratoconus or Irregular Astigmatism
Brief Title: Wavefront Guided Scleral Lenses for Keratoconus and Irregular Astigmatism
Acronym: WFG Sclerals
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cornea and Laser Eye Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLEI WFG Scleral Lens
Record Dates: First submitted 2020-12-31; First posted 2021-01-07 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Keratoconus; Irregular Astigmatism; Corneal Ectasia; Aberration, Corneal Wavefront; Wavefront Aberration, Corneal; Pellucid Marginal Corneal Degeneration; Keratoglobus
Keywords: Scleral lenses; Scleral lens; Wavefront guided scleral lenses; Higher order aberrations; HOA scleral lenses; Sclerals; Higher order aberration correction; Custom scleral lenses; Wavefront guided; Keratoconus; Irregular Astigmatism; WFG scleral lenses
MeSH Terms: conditions — Keratoconus; Corneal Wavefront Aberration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- WFG Scleral Lenses (Active Comparator): Scleral lenses with customized wavefront guided optics
  Interventions: Device: Wavefront Guided Scleral Lenses
- Traditional Scleral Lenses (Placebo Comparator): Scleral lenses with traditional optics
  Interventions: Device: Traditional Scleral Lenses

INTERVENTIONS:
Device: Wavefront Guided Scleral Lenses — Custom wavefront guided, higher order aberration correcting scleral lenses
  Other Names: ARES Scleral Lenses
  Arms: WFG Scleral Lenses
Device: Traditional Scleral Lenses — Traditional scleral lenses
  Other Names: CS Scleral Lenses
  Arms: Traditional Scleral Lenses

SUMMARY:
Aberrations are the spreading of light from a point focus. Aberrations of the eyes can be objectively evaluated with a wavefront aberrometer. Lower order aberrations such as defocus and astigmatism can be corrected with glasses and traditional/disposable soft contact lenses. Patients with ectatic corneal disease, such as keratoconus, or irregular astigmatism cause by surgery, trauma or disease, experience vision that is unlikely to be adequately corrected with glasses or disposable soft contact lenses due to higher order aberrations (HOA). HOA's cause halos, flare, glare, starbursts, doubling, smearing or ghosting of vision. Specialty contact lenses, such as scleral lenses, can be used to mask the irregularity of the cornea, reducing HOA's and improving vision. In many patients the resultant vision, though improved, still has some level of residual HOA's affecting the quality of vision. Custom scleral lenses with customized wavefront guided optics can be used to reduce residual HOA's and improve vision further. These lenses have been referred to as higher order aberration correcting scleral lenses or HOA correcting sclerals and wavefront guided scleral lenses or WFG sclerals.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the effect of an advanced technique for designing custom scleral contact lenses to further improve vision in keratoconus or irregular astigmatism by reducing residual aberrations. The derived custom scleral lenses will include customized aberration correcting optics, guided by a wavefront aberrometer measurements. These lenses are custom made based on the individual measurements from an eye.The primary objective of this study is to evaluate the vision differences between traditional scleral lens optics and customized scleral lens optics. In particular, the investigators will compare efficacy in reducing aberrations and improvement in vision.

ELIGIBILITY:
Inclusion Criteria:

-A diagnosis of keratoconus or irregular astigmatism

Exclusion Criteria:

* Patients with other visually significant ocular pathology.
* Inability to apply or remove a scleral lens.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Higher order aberration | 4 weeks
  Total higher order aberrations with traditional scleral lenses will be compared with wavefront guided scleral lenses for all eyes. A secondary analysis of this endpoint, the change in total higher order aberrations with wavefront guided scleral lenses from dispense to 4 week follow up, will be evaluated.

SECONDARY OUTCOMES:
Visual Acuity | 4 weeks
  Visual acuity with traditional scleral lenses will be compared to visual acuity with wavefront guided scleral lenses for all eyes. A secondary analysis of this endpoint, the change in visual acuity from dispense to 4 week follow up, will be evaluated for signs of neural adaptation.
Contrast Sensitivity | 4 weeks
  Contrast sensitivity with traditional scleral lenses will be compared to contrast sensitivity with wavefront guided scleral lenses for all eyes. A secondary analysis of this endpoint, the change in contrast sensitivity with wavefront guided scleral lenses from dispense to 4 week follow up, will be evaluated for signs of neural adaptation.

CONTACTS AND LOCATIONS:
Overall Officials: John D Gelles, OD, Principal Investigator — The Cornea and Laser Eye Institute
Locations (1):
- Cornea and Laser Eye Institue - Hersh Vision Group, Teaneck, New Jersey, United States